CLINICAL TRIAL: NCT03251677
Title: A Prospective Randomized Study Comparing Total Laparoscopic Hysterectomy (Lap Hysterectomy) vs Minilaparotomy (Mini-lap Hysterectomy) for Benign Uterine Lesions: Peri-operative Outcome
Brief Title: Total Laparoscopic Hysterectomy vs Minilap Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Tarek Shokeir, Prof. Obstetrics & Gynecology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD/16.12.51
Record Dates: First submitted 2017-08-10; First posted 2017-08-16 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Hysteromyoma
MeSH Terms: interventions — Surgical Procedures, Operative; Hysterectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total laparo hysterectomy (Active Comparator): Surgical procedure, Hysterectomy (removal of the uterus by laparoscopy)
  Interventions: Procedure: Surgical procedure, Hysterectomy
- Mini-lap hysterectomy (Active Comparator): Surgical procedure, Hysterectomy (removal of the uterus by mini-laparotomy)
  Interventions: Procedure: Surgical procedure, Hysterectomy

INTERVENTIONS:
Procedure: Surgical procedure, Hysterectomy — Surgical removal of the uterus

SUMMARY:
The objective of this study is to compare the perioperative outcomes between mini-lap hysterectomy and total laparoscopic hysterectomy (TLH) because of benign indications.

DETAILED DESCRIPTION:
A prospective randomized open-label study was conducted. Women >18 years of age undergoing TLH because of benign indications were recruited. Patients were randomized for either TLH (Group I, 40 cases) or minilap hysterectomy (Group II, 40 cases) through 4-5cm abdominal Pfannenstiel incision.

Inclusion criteria were mobile uterus with benign lesion and with a size up to 12 weeks gestation. Exclusion criteria adopted were patients with enlarged uterus < 12 weeks, suspected malignancy and large adnexal masses (>5cm). Peri-operative outcomes were compared.

Written informed consent was obtained from all the patients and the Departmental Ethical Committee approved the study. Patients from OB/GYN Mansoura University Hospital were enrolled. All the operations were performed by at least one of the consultants included as authors in this study.

ELIGIBILITY:
Inclusion Criteria:

* Mobile uterus.
* Uterine size up to 12 weeks gestation.
* Benign lesions.

Exclusion Criteria:

* Enlarged uterus > 12 weeks gestation.
* Suspected malignancy.
* Large adnexal masses.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Operative Time (min) | Intraoperative (Starting with induction of anesthesia (Time 0) up to complete removal of the uterus)
  Time in minutes taken for total hysterectomy
Estimated blood loss (mL) | Through surgical intervention completion
  Drop of hemoglobin and hematocrit percentage (%) 24-hours from basal pre-operative values

SECONDARY OUTCOMES:
Early postoperative complications | Within 30 days after operation
  Related complications

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Shokeir, Principal Investigator — Mansoura University
Locations (1):
- Tarek Shokeir, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Sharing up to scientific publication of a manuscript
Supporting Information: Study Protocol, CSR
Time Frame: Up to scientific publication of a manuscript
Access Criteria: Personal
URL: http://tarek.shokeir@gmail.com